CLINICAL TRIAL: NCT02768909
Title: Diagnostic Trial to Validate the Use of the E-Nose in Pulmonary TB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad Central de Venezuela (Other)
Collaborators: The ENose Company, Zutphen, Netherlands (Unknown); Foundation for Research in Mycobacteria (FUNDAIM) (Other)
Responsible Party: Principal Investigator, Jacobus H. de Waard, Chief of Tuberculosis Laboratory, Universidad Central de Venezuela
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: EN001
Record Dates: First submitted 2016-04-11; First posted 2016-05-11 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Tuberculosis, Pulmonary; e-Nose
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Electronic Nose; Surveys and Questionnaires; Restraint, Physical; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pulmonary TB (Experimental): This arm will enroll 100 patients older than 15 years old, from Caracas, with pulmonary TB, culture proved.
  Intervention:
  1. They will be asked to perform a respiration for 5 minutes through the E-Nose Device, with a nose clamp.
  2. Medical History: Symptom based Survey, Physical Exam, Anthropometric measurement.
  3. Chest X-ray.
  4. Sputum samples for Ziehl Neelsen smear and Culture in L-J.
  5. Follow Up 5 days after beginning of Tx
  6. Follow Up 15 days after beginning of Tx
  7. Follow Up 30 days after beginning of Tx
  8. Follow Up 60 days after beginning of Tx
  Interventions: Device: E-Nose; Other: Survey & Physical Exam; Other: Chest X-ray; Other: Sputum Samples; Device: Follow Up 5 days after beginning of Tx.; Device: Follow Up 15 days after beginning of Tx.; Device: Follow Up 30 days after beginning of Tx.; Device: Follow Up 60 days after beginning of Tx.
- Non - Pulmonary TB (Active Comparator): This arm will enroll 75 patients older than 15 years old, from Caracas, with non TB pulmonary infections, culture negative.
  Intervention:
  1. They will be asked to perform a respiration for 5 minutes through the E-Nose Device, with a nose clamp.
  2. Medical History: Symptom based Survey, Physical Exam, Anthropometric measurement.
  3. Chest X-ray.
  4. Sputum samples for Ziehl Neelsen smear and Culture in L-J.
  Interventions: Device: E-Nose; Other: Survey & Physical Exam; Other: Chest X-ray; Other: Sputum Samples
- Healthy Individuals (Active Comparator): This arm will enroll 75 patients older than 15 years old, from Caracas, without any symptom or sign of lower track infection.
  Intervention:
  1. They will be asked to perform a respiration for 5 minutes through the E-Nose Device, with a nose clamp.
  2. Medical History: Symptom based Survey, Physical Exam, Anthropometric measurement.
  3. Chest X-ray.
  4. Sputum samples for Ziehl Neelsen smear and Culture in L-J.
  Interventions: Device: E-Nose; Other: Survey & Physical Exam; Other: Chest X-ray; Other: Sputum Samples

INTERVENTIONS:
Device: E-Nose — 1.They will be asked to perform a respiration for 5 minutes trough the E-Nose Device, with a nose clamp.
Other: Survey & Physical Exam — 2. Perform a oriented survey for risk factors and a complete physical exam.
Other: Chest X-ray — Perform anteroposterior chest X-ray
Other: Sputum Samples — Sputum samples for Ziehl Neelsen smear and Culture in L-J.
Device: Follow Up 5 days after beginning of Tx. — Patients will be asked to come 5 days after initiation of treatment, to perform another measurement with the device.
  Also will perform a Medical History, including Symptom based Survey, Physical Exam, Anthropometric measurement, to determine progress of treatment.
  Arms: Pulmonary TB
Device: Follow Up 15 days after beginning of Tx. — Patients will be asked to come 15 days after initiation of treatment, to perform another measurement with the device.
  Also will perform a Medical History, including Symptom based Survey, Physical Exam, Anthropometric measurement, to determine progress of treatment.
  Arms: Pulmonary TB
Device: Follow Up 30 days after beginning of Tx. — Patients will be asked to come 30 days after initiation of treatment, to perform another measurement with the device.
  Also will perform a Medical History, including Symptom based Survey, Physical Exam, Anthropometric measurement, to determine progress of treatment.
  Arms: Pulmonary TB
Device: Follow Up 60 days after beginning of Tx. — Patients will be asked to come 60 days after initiation of treatment, to perform another measurement with the device.
  Also will perform a Medical History, including Symptom based Survey, Physical Exam, Anthropometric measurement, to determine progress of treatment.
  Arms: Pulmonary TB

SUMMARY:
Determine the diagnostic accuracy for pulmonary tuberculosis in adults of the E-Nose in Venezuela.

DETAILED DESCRIPTION:
Acronyms:

Tuberculosis (TB) Receiver Operating Curve (ROC) Common Terminology Criteria for Adverse Effects (CTCAE)

The aim of the study is to determine the diagnostic utility of the device 'Electronic Nose' for Pulmonary Tuberculosis. Prospective, Open, Three - Arm Controlled trial Study. Validation of the E-nose in urban settings to estimate the diagnostic accuracy of the E-nose using exhaled air in patients with Pulmonary TB in adults.

The patients who qualified for the study, according to the inclusion criteria, after consenting, will be guided through and oriented survey for risk factors, then a complete physical exam, and after that, the patient will breathe for 5 minutes trough the device, which stores the patient information, that later will be download to a computer and will be send to the server's manufacturer company, in Netherlands.

During and after the use of the device, we determine the adverse effects of the intervention, according to the CTCEA.

The researchers use the sputum culture, which is the gold standard, to determine the diagnostic utility of the test. And, will compare the results with other tests currently perform as the regular diagnostic routine, such as Chest X-ray, sputum smear, and symptom based diagnosis.

The patients in the experimental group are invited to come during the treatment phase, and will be asses the progress of the treatment, as well as another use of the device, at 5, 15, 30, 60 days after initiation of treatment, and will be compared the results of the device, with symptoms, x-ray changes, improvement of anthropometric findings, to determine the utility of the device to measure the response to treatment.

Patient Registries will be keep in an electronic database, as well as handwriting history, with the backup copy in the records of the hospital in which the patient was admitted.

auditoriae will be realised by the Ethics Comite in different time frames.

ELIGIBILITY:
Inclusion Criteria:

* Accept to participate in the study through a signed informed consent approved by the Ethical Committee of our Institution.
* More than 15 years old.
* People with a culture positive for pulmonary TB

Exclusion Criteria:

* Severe compromise of the general condition.
* Not capable to exhaled through the E-nose.
* No possibility to follow-up.
* By discretion of the research team.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of the electronic nose signal value to differentiate patients with Pulmonary TB. | 1 year
  Sensitivity, Specificity and Predictive Values; calculated with an ROC curve based on the Average processed-signal of the three electronic nose sensors. The signal is generated with a complex pattern recognition software, measuring the adsorption rate, desorption rate, and area under the curve generated by each sensor, expressed with a single value that ranges between -1 to +1.
Average Days needed to observed a negative result with the device after initiation of treatment. | 60 days
  Days-to-negative.

SECONDARY OUTCOMES:
Number of Adverse Effects related to the used of the device, assess by the CTCAE | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jacobus De Waard, PhD, Principal Investigator — Instituto de Biomedicina de la Universidad Central de Venezuela
Locations (1):
- Instituto de Biomedicina, Caracas, DC, Venezuela

IPD SHARING:
Plan to Share IPD: No